CLINICAL TRIAL: NCT03311685
Title: Vaginal Elasticity Assessment Before and After the Affect of Surgical Repair for Pelvic Organ Prolapse (POP) on Vaginal Elasticity as Measured by Vaginal Tactile Imaging
Brief Title: Vaginal Tactile Imaging for the Assessment of Pelvic Organ Prolapse Repair Efficiency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, ROY LAUTERBACH MD, Principal Investigator, Rambam Health Care Campus
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 0295-17-RMB
Record Dates: First submitted 2017-09-29; First posted 2017-10-17 (Actual); Last update posted 2020-07-27 (Actual); Status verified 2020-07

CONDITIONS: Pelvic Organ Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laparoscopic POP repair (Experimental): Patients undergoing laparoscopic surgery for the repair of pelvic organ prolapse.
  vaginal tactile imager
  Interventions: Device: vaginal tactile imager
- Vaginal POP repair (Experimental): Patients undergoing vaginal surgery for the repair of pelvic organ prolapse. vaginal tactile imager
  Interventions: Device: vaginal tactile imager

INTERVENTIONS:
Device: vaginal tactile imager — Patients will undergo elasticity assessment with vaginal tactile imaging the be once before surgical repair and twice after surgery in a 3 month interval.

SUMMARY:
Female patients with POP will be evaluated for vaginal elasticity using vaginal tactile imaging both before and after surgery for the repair of the POP. Surgical repair will be performed by a single surgeon who will perform either a laparoscopic or vaginal repair.

DETAILED DESCRIPTION:
Patients will be recruited and sign a consent form. The patients included are patients with POP that are candidates for either laparoscopic or vaginal repair.

Assessment of vaginal elasticity via vaginal tactile imaging will be performed at 3 different points:

* The day of surgery before surgery.
* The day after surgery.
* 3 months post-operational. Every patient will serve as her own control. Demographic, gynecologic and obstetric history will be obtained from patients' electronic files.

ELIGIBILITY:
Inclusion Criteria:

* Any woman undergoing POP repair

Exclusion Criteria:

* Women above or below the age limit

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 30 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-07-20 (Actual)

PRIMARY OUTCOMES:
Vaginal elasticity assessment | Up to 3 months from enrollment
  Vaginal elasticity as measured by the vaginal tactile imager measuring the local vaginal pressure (in mmHg)

SECONDARY OUTCOMES:
Comparison of vaginal elasticity between repair methods | Up to 3 months from enrollment
  Assessment of the difference in vaginal elasticity (measured in mmHg) between the laparoscopic and vaginal surgical repair groups.

CONTACTS AND LOCATIONS:
Overall Officials: Roy Lauterbach, MD, Principal Investigator — Rambam healthcare campus
Locations (1):
- Rambam health care campus, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No